CLINICAL TRIAL: NCT06590701
Title: Scapholunate Ligament Reconstruction: Early Dart Throwing Motion Versus Motion in Anatomical Planes
Acronym: SL-Reko
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Reissner (Other)
Responsible Party: Sponsor-Investigator, Lisa Reissner, Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-Reko
Record Dates: First submitted 2024-05-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Scapholunate Ligament Rupture
Keywords: Mobilisation; Scapholunate ligament recontruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early dart throwing motion (Experimental): From the 2nd postoperative week, the 'Dart-Throwing Motion' is started, from radial extension to ulnar flexion.
  Interventions: Other: Early dart throwing motion-mobilization
- Mobilisation in anatomical planes (Active Comparator): From the 2nd postoperative week, movements are started in the anatomical plane of the hand (standard rehabilitation)
  Interventions: Other: Early dart throwing motion-mobilization

INTERVENTIONS:
Other: Early dart throwing motion-mobilization — We compare two different mobilisations in the rehabilitation of patients following scapholunate ligament reconstruction

SUMMARY:
Patients undergoing scapholunate ligament reconstruction at Balgrist University Hospital are divided into two groups and receive two different types of mobilisation postoperatively. The investigators will compare the outcome (pain, strength, mobility) between the two groups 1 year after the operation.

DETAILED DESCRIPTION:
The so-called 'dart-throwing motion' (DTM) plane of movement, from radial extension to ulnar flexion, has gained attention as it has been shown to be an important axis of wrist movement during activities of daily living. Further studies have shown that during movement of the intact wrist in the dart throwing plane, most of the movement occurs in the mediocarpal joint, while the proximal row remains relatively immobile.

In scapholunate (SL) ligament reconstruction using the flexor carpi radialis tendon, the SL interval is immobilised using 2 Kirschner wires for 8-10 weeks to relieve the strain on the ligament and allow it to heal. From the 2nd postoperative week, mobilisation is started using DTM mobilisation or mobilisation in the anatomical plane. The aim of the study is to investigate in a randomised trial whether mobilisation in the anatomical plane produces the same postoperative results.

In this project, the investigators will compare two types of mobilisation in the rehabilitation of SL ligament reconstruction. The participants will be randomised to two treatment groups. This procedure therefore corresponds to a risk category A in 'other' clinical trials according to Chapter 4 ClinO.

ELIGIBILITY:
Inclusion Criteria:

* SL Ligament reconstruction at Balgrist University Hospital
* at least 18 years
* Written informed consent

Exclusion Criteria:

* Age under 18 years
* Refusal of participation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain in resting position | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of resting pain using the VAS Score (Visual Analog Scale), where 0 indicates no pain and 10 indicates the worst pain.
Pain during activity | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of pain during activity using the VAS (Visual Analog Scale), where 0 indicates no pain and 10 indicates the worst pain
Mobility of the wrist: Flexion | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of wrist flexion by measuring the range of motion in degrees.
Mobility of the wrist: Extension | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of wrist extension by measuring the range of motion in degrees.
Mobility of the wrist: Ulnar deviation | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of wrist ulnar deviation by measuring the range of motion in degrees.
Mobility of the wrist: Pronation | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of wrist pronation by measuring the range of motion in degrees.
Mobility of the wrist: Supination | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Assessment of wrist supination by measuring the range of motion in degrees.
Strength Assessment: Grip Strength | Before surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Using the Jamar Hydraulic Hand Dynamometer which displays isometric grip force from 0-90 kg, grip strength will be assessed.

SECONDARY OUTCOMES:
Recording ability to work | Before surgery, 7 weeks after surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Degree of employment in per cent (from 0 to a maximum of 100 per cent) is recorded
Recording of physical limitations | Before surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Using the DASH (Disabilities of the Arm, Shoulder, and Hand) questionnaire, physical limitation will be recorded. This 30-item questionnaire allows patients to rate difficulty and interference with daily life on a 5-point Likert scale. The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Recording wrist pain and restrictions | Before surgery, 11 weeks after surgery, 6 months after surgery, 12 months after surgery
  Using the PRWE (Patient-Rated Wrist Evaluation) questionnaire, specific wrist pain and restrictions will be recorded. This 15-item questionnaire measures wrist pain and disability in daily activities. Patients rate their wrist pain and disability from 0 (no pain) to 10 (worst pain).
  * Pain subscale:Contains 5 items, each rated from 0 to 10, with a maximum score of 50 and a minimum of 0.
  * Function subscale: Contains 10 items divided into two sections: specific activities (6 items) and usual activities (4 items). The maximum score is 50 and the minimum is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Reissner, PD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crisco JJ, Wilcox BJ, Beckwith JG, Chu JJ, Duhaime AC, Rowson S, Duma SM, Maerlender AC, McAllister TW, Greenwald RM. Head impact exposure in collegiate football players. J Biomech. 2011 Oct 13;44(15):2673-8. doi: 10.1016/j.jbiomech.2011.08.003. Epub 2011 Aug 27. PMID 21872862
- [Background] Werner FW, Green JK, Short WH, Masaoka S. Scaphoid and lunate motion during a wrist dart throw motion. J Hand Surg Am. 2004 May;29(3):418-22. doi: 10.1016/j.jhsa.2004.01.018. PMID 15140483
- [Background] Crisco JJ, Coburn JC, Moore DC, Akelman E, Weiss AC, Wolfe SW. In vivo radiocarpal kinematics and the dart thrower's motion. J Bone Joint Surg Am. 2005 Dec;87(12):2729-2740. doi: 10.2106/JBJS.D.03058. PMID 16322624
- [Background] Moritomo H, Apergis EP, Herzberg G, Werner FW, Wolfe SW, Garcia-Elias M. 2007 IFSSH committee report of wrist biomechanics committee: biomechanics of the so-called dart-throwing motion of the wrist. J Hand Surg Am. 2007 Nov;32(9):1447-53. doi: 10.1016/j.jhsa.2007.08.014. PMID 17996783